CLINICAL TRIAL: NCT03466346
Title: A Sequential, Multiple Assignment Randomized Trial (SMART) for Non-specialist Treatment of Common Mental Disorders in Kenya: Leveraging the Depression And Primary-care Partnership for Effectiveness-implementation Research (DAPPER) Project
Brief Title: SMART-DAPPER: Leveraging the Depression And Primary-care Partnership for Effectiveness-implementation Research Project
Acronym: SMART-DAPPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Nairobi (Other); National Institute of Mental Health (NIMH) (NIH); Kenya Medical Research Institute (Other); University of California, San Diego (Other); Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R01MH115512 1R01MH113722-01A1; 1R01MH115512 (NIH); 1R01MH113722-01A1 (NIH)
Record Dates: First submitted 2018-03-02; First posted 2018-03-15 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Depression, Unipolar; Posttraumatic Stress Disorder; Trauma
MeSH Terms: conditions — Depressive Disorder; Stress Disorders, Post-Traumatic; Wounds and Injuries | interventions — Fluoxetine; Interpersonal Psychotherapy

STUDY DESIGN:
Intervention Model Description: fluoxetine versus interpersonal psychotherapy (IPT) for treatment of Major Depressive Disorder (MDD) and/or Posttraumatic Stress Disorder (PTSD)
Who Masked: Outcomes Assessor
Masking Description: participants will be evaluated by an outcomes assessor that is not aware of which treatment the participant is receiving. This will be achieved by keeping the randomization key locked and accessible only to the study coordinator and investigators. Participants who are scheduled for assessments will be reminded not to spontaneously disclose their treatment modality to the outcomes assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Interpersonal psychotherapy (Active Comparator): IPT was developed in the 1980s by Gerald Klerman and Myrna Weissman to address interpersonal issues in depression. IPT is now considered evidence-based, first-line treatment for depression. IPT improves symptoms by addressing problems in social relationships. IPT is traditionally delivered as weekly one-hour sessions over 12 weeks, focused on one interpersonal problem area.
  Interventions: Behavioral: Interpersonal Psychotherapy
- fluoxetine (Active Comparator): Fluoxetine is a selective serotonin reuptake inhibitor that is FDA approved for the treatment of depression. Compared to placebo, fluoxetine is more likely to produce symptom response for MDD. Despite the interim development of many other antidepressants since the development of fluoxetine, it remains a first line treatment for depression.
  Interventions: Drug: Fluoxetine
- Fluoxetine after IPT (Active Comparator): participants who do not remit from MDD and PTSD after treatment with IPT may be randomized to fluoxetine.
  Interventions: Drug: Fluoxetine
- IPT after fluoxetine (Active Comparator): participants who do not remit from MDD and PTSD after treatment with fluoxetine may be randomized to IPT.
  Interventions: Behavioral: Interpersonal Psychotherapy
- IPT + fluoxetine (Active Comparator): participants who do not remit from MDD and PTSD after treatment with fluoxetine may be randomized to IPT + fluoxetine.
  Interventions: Drug: Fluoxetine; Behavioral: Interpersonal Psychotherapy

INTERVENTIONS:
Drug: Fluoxetine — Fluoxetine is a selective serotonin reuptake inhibitor that is FDA approved for the treatment of depression. Compared to placebo, fluoxetine is more likely to produce symptom response for MDD. Despite the interim development of many other antidepressants since the development of fluoxetine, it remains a first line treatment for depression.
  Arms: Fluoxetine after IPT; IPT + fluoxetine; fluoxetine
Behavioral: Interpersonal Psychotherapy — IPT was developed in the 1980s by Gerald Klerman and Myrna Weissman to address interpersonal issues in depression. IPT is now considered evidence-based, first-line treatment for depression. IPT improves symptoms by addressing problems in social relationships. IPT is traditionally delivered as weekly one-hour sessions over 12 weeks, focused on one interpersonal problem area.
  Other Names: IPT
  Arms: IPT + fluoxetine; IPT after fluoxetine; Interpersonal psychotherapy

SUMMARY:
Despite carrying the vast majority of the global mental disorder burden, 75% of adults with mental disorders in Low and Middle Income Countries have no access to services. This study will test strategies for integrating first and second line evidence-based depression and trauma-related disorder treatments with primary care services at a large public sector hospital and conduct robust cost and cost-benefit analyses of each treatment to produce a "menu" of cost-benefit options for personalized, integrated mental health care with corresponding effectiveness and implementation values.

DETAILED DESCRIPTION:
Mental disorders are a leading cause of global disability, driven by depression and anxiety. Most of the disease burden is in Low and Middle Income Countries (LMICs), where 75% of adults with mental disorders have no service access. Despite nearly 15 years of efficacy research showing that local non-specialists can provide evidence-based care for depression and anxiety in LMICs, few studies have advanced to the critical next step: identifying strategies for sustainable "real world" non-specialist treatment including integration with existing healthcare platforms and response to common clinical dilemmas, such as what treatment to start with and how to modify it.

Given the need to personalize treatment to achieve remission (absence of disease) and the scarcity of mental health specialists in LMICs, successful reduction of population-level disability caused by depression and anxiety requires (1) evidence-based strategies for first-line and second-line (non-remitter) treatment delivered by non-specialists, with (2) confirmation of presumed mechanism of action and (3) patient-level moderators of treatment outcome to inform personalized, non-specialist treatment algorithms.

The research team has worked in western Kenya for 6 years with a UCSF-Kenya collaboration that supports integrated HIV services at over 70 primary healthcare facilities in Kisumu County (Family AIDS Care and Education Services [FACES]). Primary care populations in Kenya have high prevalence of Major Depressive Disorder (MDD) (26%) and Posttraumatic Stress Disorder (PTSD) (35%). Kenyan leaders lack an evidence base for two essential treatments - psychotherapy and second generation antidepressants- without which scale-up will fall short of its potential. We conducted a randomized, controlled trial in Kisumu County of Interpersonal Psychotherapy (IPT) delivered by non-specialists for HIV-positive patients with MDD and PTSD. In our study, IPT achieved full remission of MDD and PTSD in the majority of participants.

Given the high prevalence of MDD-PTSD co-morbidity, we will collaborate with the FACES team providing services to Kisumu County Hospital (KCH) primary care outpatient clinic (~10,000 patients/month) to conduct a randomized trial of IPT versus fluoxetine for MDD and/or PTSD. Local non-specialists will be trained in mental health care for the SMART and hired through the Kenyan Ministry of Health to work at KCH. SMART participants will be randomized to: (1) first line treatment with IPT or fluoxetine; (2) second line treatment for non-remitters- treatment "switch" (e.g., IPT to fluoxetine) or treatment "combination" (e.g., addition of IPT to fluoxetine). Research with mental health specialists in high income countries suggests that antidepressants and psychotherapy have equivalent short-term efficacy and that psychotherapy yields superior long-term relapse prevention. We will test the role of previously identified mechanisms in mediating remission and key moderators of treatment effect. Results of moderator and Q learning analyses will produce first and second-line non-specialist treatment algorithms.

ELIGIBILITY:
Inclusion Criteria:

1. Kisumu County Hospital (KCH) adult primary care outpatient clinic attendees who screen positive for depression and/or PTSD
2. Ability to attend weekly IPT sessions/fluoxetine monitoring; (3) 18 years or older

Exclusion Criteria:

1. Cognitive dysfunction compromising ability to participate in IPT or accurately take fluoxetine (lack of orientation to person, place, time and situation)
2. acute suicidality requiring higher level of care
3. drug/alcohol use disorders requiring substance use treatment (AUDIT score of 8 or higher, DAST score of 3 or higher)
4. history of mania or requiring treatment for hypomania
5. Outside mental health treatment during the study treatment phases (any mental health treatment is allowed during follow-up phases and is recorded by study team).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2162 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muthoni J Mathai, MDChB, MMed, Principal Investigator — University of Nairobi; Susan M Meffert, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (3):
- Kenya (3):
  - Jaramogi Oginga Odinga Teaching and Referral Hospital (JOOTRH), Kisumu
  - Kisumu County Hospital, Kisumu
  - Lumumba Health Center, Kisumu

IPD SHARING:
Plan to Share IPD: Yes
NIMH Data Archive The National Institutes of Health (NIH) and NIMH have developed a federation of data repositories called the NIMH Data Archive (NDA) to store the collection of data from participants in research studies related to mental health, regardless of the source of funding. The extensive information collected by these studies, and subsequently stored in the National Database for Autism Research (NDAR), the NIH Pediatric MRI Repository (PedsMRI), the National Database for Clinical Trials Related to Mental Illness (NDCT), and the Research Domain Criteria Database (RDoCdb) provides a rare and valuable scientific resource. The NIH and the NIMH seek to encourage the use of these resources to achieve rapid scientific progress. In order to take full advantage of such resources and maximize their research value, it is important that data be made available, on appropriate terms and conditions, to the largest possible number of qualified investigators in a timely manner.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be made available to the NIMH data archive as soon as it is verified as clean and complete, with at least annual updates throughout the duration of the study. Data will be be available indefinitely or for as long as the NIMH repositories supports the electronic data storage.
Access Criteria: The investigative team and our NIMH and GACD partners will review requests for data. Evaluation will include scientific merit of the proposal, overlap versus building upon the study goals.

REFERENCES:
- [Derived] Mwai D, Meffert SM, Olwanda EE, Mathai MA, Ongeri L, Burger RL, Mbwayo A, Rota G, Otieno A, Cohen CR, Bukusi D, Aarons GA, Neylan TC, McCulloch CE, Jin C, Akena D, Kahonge S, Kahn JG. Productivity benefits of treatment of depression and post-traumatic stress disorder in Kenya. BMJ Glob Health. 2025 Nov 3;10(11):e018204. doi: 10.1136/bmjgh-2024-018204. PMID 41184028
- [Derived] Burger RL, Meffert SM meffert, Ongeri L, Wangia J, Wambura R, Ajore P, Rota G, Otieno A, Obura RR, Muchembre P, Bukusi D, Mbwayo A, Neylan TC, Akena D, Jin C, McCulloch C, Mathai MA. Factors associated with fluoxetine adherence among outpatients with common mental disorders in Western Kenya. BMJ Glob Health. 2025 Aug 25;10(8):e017929. doi: 10.1136/bmjgh-2024-017929. PMID 40854809
- [Derived] Olwanda E, Mwai D, Mathai M, Burger R, Ongeri L, Bukusi D, Mbwayo A, Rota G, Otieno A, Rota R, Meffert S, Kahn JG. Cost-Benefit Analysis of Interpersonal Therapy and Fluoxetine for Treating Depression and PTSD in Primary Care Settings in Kenya. Res Sq [Preprint]. 2025 Jul 28:rs.3.rs-6977800. doi: 10.21203/rs.3.rs-6977800/v1. PMID 40766223
- [Derived] Meffert S, Mathai M, Neylan T, Mwai D, Onyango DO, Rota G, Otieno A, Obura RR, Wangia J, Opiyo E, Muchembre P, Oluoch D, Wambura R, Mbwayo A, Kahn JG, Cohen CR, Bukusi D, Aarons GA, Burger RL, Jin C, McCulloch C, Kahonge S, Ongeri L. Preference of mHealth versus in-person treatment for depression and post-traumatic stress disorder in Kenya: demographic and clinical characteristics. BMJ Open. 2024 Nov 18;14(11):e083094. doi: 10.1136/bmjopen-2023-083094. PMID 39557549
- [Derived] Getahun M, Mathai MA, Rota G, Allen A, Burger RL, Opiyo E, Oluoch D, Wangia J, Wambura R, Mbwayo A, Muchembre P, Obura RR, Neylan TC, Aarons GA, Ongeri L, Meffert SM. "The peace that I wanted, I got": Qualitative insights from patient experiences of SMART DAPPER interventions for major depression and traumatic stress disorders in Kenya. PLOS Glob Public Health. 2024 Sep 5;4(9):e0002685. doi: 10.1371/journal.pgph.0002685. eCollection 2024. PMID 39236052
- [Derived] Levy R, Mathai M, Chatterjee P, Ongeri L, Njuguna S, Onyango D, Akena D, Rota G, Otieno A, Neylan TC, Lukwata H, Kahn JG, Cohen CR, Bukusi D, Aarons GA, Burger R, Blum K, Nahum-Shani I, McCulloch CE, Meffert SM. Implementation research for public sector mental health care scale-up (SMART-DAPPER): a sequential multiple, assignment randomized trial (SMART) of non-specialist-delivered psychotherapy and/or medication for major depressive disorder and posttraumatic stress disorder (DAPPER) integrated with outpatient care clinics at a county hospital in Kenya. BMC Psychiatry. 2019 Dec 28;19(1):424. doi: 10.1186/s12888-019-2395-x. PMID 31883526

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: N=1682 Screened Out for =>1 reason/ppt
  * 384 Didn't return -956 MDE- & PTSD-
  * 179 Drug or Alcohol Use
  * 120 Suicidality
  * 100 Unwilling to ppt
  * 133 History/Current Mania
  * 82 Pregnant or Breastfeeding
  * 13 Taking FLX
  * 1 Age <18
  * 2 Didn't consent
  * 2 Current ppt
  * 6 Cognitive dysfunction
  N= 20 Eligible and Not Randomized for =>1 reason/ppt
  * 6 Declined
  * 7 Specialized or Higher level of care
  * 2 Moved out
  * 2 Pregnant or breastfeeding
  * 2 Drug or Alcohol Use
  * 1 Boarding school
Groups:
- Stage 1: Interpersonal Psychotherapy: IPT was developed in the 1980s by Gerald Klerman and Myrna Weissman to address interpersonal issues in depression. IPT is now considered evidence-based, first-line treatment for depression. IPT improves symptoms by addressing problems in social relationships. IPT is traditionally delivered as weekly one-hour sessions over 12 weeks, focused on one interpersonal problem area.
  Interpersonal Psychotherapy: IPT was developed in the 1980s by Gerald Klerman and Myrna Weissman to address interpersonal issues in depression. IPT is now considered evidence-based, first-line treatment for depression. IPT improves symptoms by addressing problems in social relationships. IPT is traditionally delivered as weekly one-hour sessions over 12 weeks, focused on one interpersonal problem area.
- Stage 1: Fluoxetine: Fluoxetine is a selective serotonin reuptake inhibitor that is FDA approved for the treatment of depression. Compared to placebo, fluoxetine is more likely to produce symptom response for MDD. Despite the interim development of many other antidepressants since the development of fluoxetine, it remains a first line treatment for depression.
  Fluoxetine: Fluoxetine is a selective serotonin reuptake inhibitor that is FDA approved for the treatment of depression. Compared to placebo, fluoxetine is more likely to produce symptom response for MDD. Despite the interim development of many other antidepressants since the development of fluoxetine, it remains a first line treatment for depression.
- Stage 2: IPT After Fluoxetine: Participants who did not remit with fluoxetine and were randomized to receive second line treatment with IPT
- Stage 2: Fluoxetine After IPT: Participants who did not remit with IPT and were randomized to receive second line treatment with fluoxetine.
- Stage 2: IPT and Fluoxetine: Combination treatment with both IPT and fluoxetine for participants who did not remit with IPT or fluoxetine
Period: Stage 1 - 1st Line Trt (IPT or FLX)
Arm/Group | Stage 1: Interpersonal Psychotherapy | Stage 1: Fluoxetine | Stage 2: IPT After Fluoxetine | Stage 2: Fluoxetine After IPT | Stage 2: IPT and Fluoxetine
Started | 1082 | 1080 | 0 | 0 | 0
Completed | 986 | 878 | 0 | 0 | 0
Not Completed | 96 | 202 | 0 | 0 | 0
Not completed — Death | 0 | 3 | 0 | 0 | 0
Not completed — Physician Decision | 12 | 26 | 0 | 0 | 0
Not completed — Participant withdrawal or relocated | 15 | 31 | 0 | 0 | 0
Not completed — Lost to Follow-up | 69 | 142 | 0 | 0 | 0
Period: Stage 2 - 2nd Line Trt (Combo or Switch)
Arm/Group | Stage 1: Interpersonal Psychotherapy | Stage 1: Fluoxetine | Stage 2: IPT After Fluoxetine | Stage 2: Fluoxetine After IPT | Stage 2: IPT and Fluoxetine
Started | 0 | 0 | 68 | 104 | 160
Completed | 0 | 0 | 50 | 77 | 109
Not Completed | 0 | 0 | 18 | 27 | 51
Not completed — Physician Decision | 0 | 0 | 2 | 1 | 4
Not completed — Participant withdrawal or relocated | 0 | 0 | 0 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 16 | 24 | 45

BASELINE CHARACTERISTICS:
Population: stage 2 participants do not have baseline data
Groups:
- Stage 1: Interpersonal Psychotherapy (IPT): 3 months of weekly IPT sessions
- Stage 1: Fluoxetine: 6 months of fluoxetine. Participants began with 20mg 1 tablet per day. If symptom reduction did not occur, the dose was increased by 20mg increments each month to an upper limit of 60mg.
- Stage 2: Fluoxetine After IPT: Participants who were not in remission after IPT who received second line treatment with fluoxetine
- Stage 2: IPT After Fluoxetine: Participants who were not in remission after fluoxetine who received second line treatment with IPT
- Stage 2: Fluoxetine and IPT: Participants who were not in remission after IPT or fluoxetine who received second line treatment with fluoxetine and IPT
- Total: Total of all reporting groups
Arm/Group | Stage 1: Interpersonal Psychotherapy (IPT) | Stage 1: Fluoxetine | Stage 2: Fluoxetine After IPT | Stage 2: IPT After Fluoxetine | Stage 2: Fluoxetine and IPT | Total
Number analyzed (Participants) | 1082 | 1080 | 0 | 0 | 0 | 2162
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (11.2) | 35.3 (10.8) |  |  |  | 35.7 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 977 | 981 |  |  |  | 1958
  Male | 105 | 99 |  |  |  | 204
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  |  |  | 0
  Asian | 0 | 0 |  |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  |  | 0
  Black or African American | 1082 | 1080 |  |  |  | 2162
  White | 0 | 0 |  |  |  | 0
  More than one race | 0 | 0 |  |  |  | 0
  Unknown or Not Reported | 0 | 0 |  |  |  | 0
Region of Enrollment [Number; unit: participants]
  Kenya | 1082 | 1080 |  |  |  | 2126
Major Depression on Mini International Neuropsychiatric Interview (MINI) [Count of Participants; unit: Participants] | 1035 | 1036 |  |  |  | 2071
PTSD (Mini International Neuropsychiatric Interview (MINI) [Count of Participants; unit: Participants] | 555 | 563 |  |  |  | 1118
Major Depression adn PTSD (MINI) [Count of Participants; unit: Participants] | 508 | 519 |  |  |  | 1027
Depression symptoms (BDI2) [Mean (Standard Deviation); unit: BDI2 cutscore 19 for major depressio] — Beck Depression Inventory-Second Edition (BDI-II) score of 19 or greater is defined as positive for major depression. BDI-II score below 19 is defined as negative for major depression. Scores range from 0 to 63 with higher total scores indicating more severe depressive symptoms.
  BDI2 cutscore 19 for major depressio | 28.7 (10.3) | 29.1 (10.5) |  |  |  | 28.9 (10.4)
PTSD symptoms (PCL) [Mean (Standard Deviation); unit: PCL-5 cutscore 23 for PTSD] — PTSD Checklist for DSM-5 (PCL-5) score of 23 or greater is defined as positive for PTSD. PCL-5 score below 23 is defined as negative for PTSD. Score range from 0 to 80 with higher total scores indicating more severe PTSD symptoms.
  PCL-5 cutscore 23 for PTSD | 43.6 (17.4) | 43.3 (17.2) |  |  |  | 43.5 (17.3)
HIV co-morbidity [Count of Participants; unit: Participants] | 438 | 413 |  |  |  | 851
Other co-morbidity (hypertension, diabetes, tuberculosis, syphilis, hypothyroidism, hyperthyroidism) [Count of Participants; unit: Participants] | 99 | 96 |  |  |  | 195
History of Mental Health Care [Count of Participants; unit: Participants] | 10 | 13 |  |  |  | 23
Lifetime physical intimate partner violence among partnered participants [Count of Participants; unit: Participants] — The Conflict Tactics Scale (CTS2) short form is a widely used measure of intimate partner violence (IPV). We examined the subscale for physical IPV among partnered participants. Given the high prevalence of IPV in the region, its association with depression and PTSD, and promising studies showing reduction of IPV with treatment of depression and PTSD, we evaluated IPV among partnered participants baseline and follow up. Population: Partnered participants
  Participants
    number analyzed (Participants) | 551 | 568 | 0 | 0 | 0 | 1119
    (all) | 319 | 343 |  |  |  | 662

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Depression at End of Treatment
Description: Number of Participants with Major Depression. The Beck Depression Inventory-Second Edition (BDI-II) was used and a score of 19 or greater was defined as positive for major depression. BDI-II score below 19 is defined as negative for major depression. Scores range from 0 to 63 with higher total scores indicating more severe depressive symptoms.
Time Frame: End of 1st line Treatment (up to month 6) and end of 2nd line Treatment (up to month 12)
Population: Number of participants with Major Depression in each arm at the end of 1st line Treatment (Stage 1) and the end of 2nd line Treatment (Stage 2)
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Interpersonal Psychotherapy (IPT) | Stage 1: Fluoxetine | Stage 2: Fluoxetine After IPT | Stage 2: IPT After Fluoxetine | Stage 2: Fluoxetine and IPT
Number analyzed (Participants) | 986 | 878 | 77 | 50 | 109
Participants | 127 | 89 | 6 | 11 | 11

2. Primary Outcome: Number of Participants With PTSD
Description: Number of Participants with PTSD. The PTSD Checklist for DSM-5 (PCL-5) was used and score of 23 or greater is defined as positive for PTSD. PCL-5 score below 23 is defined as negative for PTSD. Score range from 0 to 80 with higher total scores indicating more severe PTSD symptoms.
Time Frame: End of 1st line Treatment (up to month 6) and end of 2nd line Treatment (up to month 12)
Population: Number of participants with PTSD in each arm at end of 1st line Treatment (Stage 1) and end of 2nd line Treatment (Stage 2)
Measure: Count of Participants; unit: Participants
Groups:
- Stage 2: IPT After Fluoxetine: IPT After Fluoxetine - Participants who were not in remission after fluoxetine who received second line treatment with IPT
Arm/Group | Stage 1: Interpersonal Psychotherapy (IPT) | Stage 1: Fluoxetine | Stage 2: Fluoxetine After IPT | Stage 2: IPT After Fluoxetine | Stage 2: Fluoxetine and IPT
Number analyzed (Participants) | 986 | 878 | 77 | 50 | 109
Participants | 173 | 108 | 10 | 14 | 20

ADVERSE EVENTS:
Time Frame: 30 month follow-up
Groups:
- Stage 1: Interpersonal Psychotherapy (IPT): 3 months of weekly Interpersonal Psychotherapy sessions
- Stage 2: Fluoxetine and IPT: IPT or fluoxetine participants who are not in remission at the end of first line treatment who receive IPT and fluoxetine (combination) as second line treatment
Arm/Group | Stage 1: Interpersonal Psychotherapy (IPT) | Stage 1: Fluoxetine | Stage 2: IPT After Fluoxetine | Stage 2: Fluoxetine After IPT | Stage 2: Fluoxetine and IPT
All-Cause Mortality (participants affected / at risk) | 7/1082 | 14/1080 | 1/68 | 1/104 | 0/160
Serious Adverse Events (participants affected / at risk) | 37/1082 | 49/1080 | 3/68 | 6/104 | 8/160
Other Adverse Events (participants affected / at risk) | 326/1082 | 139/1080 | 5/68 | 10/104 | 16/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: Interpersonal Psychotherapy (IPT) (N=1082) | Stage 1: Fluoxetine (N=1080) | Stage 2: IPT After Fluoxetine (N=68) | Stage 2: Fluoxetine After IPT (N=104) | Stage 2: Fluoxetine and IPT (N=160)
Gastrointestinal distress (Gastrointestinal disorders) | 1 | 5 | 0 | 0 | 0 — For example diarrhea, vomiting
Ob/gyn (Reproductive system and breast disorders) | 5 | 5 | 1 | 1 | 0 — Ob/gyn events
Fatigue/Malaise (General disorders) | 1 | 0 | 0 | 0 | 0 — Fatigue/Malaise
Ear Nose and Throat (ENT) (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 — Ear Nose and Throat (ENT)
Abnormal laboratory result (Investigations) | 2 | 1 | 0 | 0 | 0 — Abnormal laboratory results
Musculoskeletal (MS) (Musculoskeletal and connective tissue disorders) | 2 | 4 | 1 | 0 | 1 — Musculoskeletal (MS)
Other SAEs (General disorders) | 4 | 13 | 0 | 2 | 0 — Other SAEs
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 — Pain
Typhoid (Infections and infestations) | 2 | 0 | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 2 | 3 | 0 | 0 | 0 — Injury
Respiratory (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 0 | 1
Malaria (Infections and infestations) | 3 | 3 | 0 | 2 | 4 — Malaria
Dysphagia / odynophagia (General disorders) | 1 | 0 | 0 | 0 | 0 — Dysphagia / odynophagia
Cardiovascular (CV) (Cardiac disorders) | 1 | 2 | 0 | 0 | 0 — Cardiovascular (CV)
Thought of self-harm or suicidal ideation (Psychiatric disorders) | 6 | 2 | 0 | 0 | 1 — Thought of self-harm or suicidal ideation
Endocrine/Metabolic (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 — Endocrine/Metabolic
Hemopoietic sysytem (Blood and lymphatic system disorders) | 1 | 2 | 1 | 0 | 0 — Hemopoietic sysytem
bacterial/fungal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 — bacterial/fungal infection
Jaundice (General disorders) | 0 | 1 | 0 | 0 | 0 — Jaundice
Neurological (Nervous system disorders) | 1 | 3 | 0 | 0 | 0 — Neurological
Renal system (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 — Renal system
Sexual dysfunction (General disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: Interpersonal Psychotherapy (IPT) (N=1082) | Stage 1: Fluoxetine (N=1080) | Stage 2: IPT After Fluoxetine (N=68) | Stage 2: Fluoxetine After IPT (N=104) | Stage 2: Fluoxetine and IPT (N=160)
Abdominal Pain (Gastrointestinal disorders) | 12 | 2 | 0 | 0 | 2
Abnormal Laboratory Results (Investigations) | 1 | 1 | 0 | 0 | 0
Thoughts of self-harm (Psychiatric disorders) | 6 | 3 | 0 | 0 | 0
Burn (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 0 | 0
Cardiovascular (Cardiac disorders) | 8 | 6 | 0 | 1 | 0
Chest pain (Cardiac disorders) | 15 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 6 | 0 | 0 | 1
Dizziness (General disorders) | 1 | 1 | 0 | 0 | 1
Ear Nose and Throat (Ear and labyrinth disorders) | 11 | 5 | 0 | 0 | 0
Endocrine/Metabolic (Endocrine disorders) | 2 | 4 | 0 | 0 | 0
Fatigue/Malaise (General disorders) | 7 | 6 | 0 | 1 | 0
Fever (General disorders) | 4 | 2 | 0 | 0 | 0
Gastrointestinal Distress (Gastrointestinal disorders) | 10 | 17 | 0 | 1 | 0
Genitourinary (GU) (Renal and urinary disorders) | 7 | 4 | 0 | 0 | 0
Headache (General disorders) | 34 | 5 | 1 | 1 | 1
Hemopoietic System (General disorders) | 1 | 4 | 0 | 0 | 0
Infection - bacterial/fungal (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 10 | 1 | 0 | 0 | 1
Jaundice (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Malaria (Infections and infestations) | 56 | 15 | 0 | 1 | 2
Miscellaneous (General disorders) | 20 | 14 | 1 | 2 | 1
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 27 | 4 | 0 | 1 | 1
Neurological (Nervous system disorders) | 3 | 1 | 0 | 0 | 0
OBGYN (Reproductive system and breast disorders) | 3 | 6 | 0 | 1 | 0
Pain (General disorders) | 34 | 6 | 0 | 0 | 1
Pallor (General disorders) | 1 | 0 | 0 | 1 | 0
Renal System (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0
Respiratory (Respiratory, thoracic and mediastinal disorders) | 25 | 8 | 1 | 0 | 5
Sedation (General disorders) | 0 | 3 | 0 | 0 | 0
Seizure (General disorders) | 0 | 2 | 0 | 0 | 0
Sexual Disfunction (General disorders) | 0 | 1 | 0 | 0 | 0
Skin (Skin and subcutaneous tissue disorders) | 7 | 5 | 0 | 0 | 0
Sweating (General disorders) | 0 | 5 | 0 | 0 | 0
Thyroid (General disorders) | 1 | 0 | 0 | 0 | 0
Typhoid (Infections and infestations) | 3 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/46/NCT03466346/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/46/NCT03466346/SAP_001.pdf